CLINICAL TRIAL: NCT02045641
Title: The Clinical Impact of an Aggressive Approach Towards Pleural and Pericardial Effusions Following Open Heart Surgery: a Step Towards Standard Guidelines
Brief Title: Pleural and Pericardial Effusion Following Open Heart Surgery
Acronym: IMAGING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Laura Sommer Hansen, MD PHD fellow, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-246-13
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Heart Disease; Pleural Effusion; Pericardial Effusion
Keywords: cardiac surgery; postoperative treatment; pleural effusion; physical performance
MeSH Terms: conditions — Heart Diseases; Pleural Effusion; Pericardial Effusion | interventions — Thoracentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- current postoperative regimen (No Intervention): The group will follow the current postoperative regimen at the surgical ward; screening for pleural effusions with x-ray and further diagnostic procedures in case of symptoms. Treatment will be entirely in the hands of the clinical personnel.
- pleuracentesis (Experimental): The group will follow the current postoperative regimen. In addition they will be followed with ultrasound examination, clinical examination, spirometry examination and 6 minute walk test. In case of either a) pleural effusion > 400ml OR b) pleural effusion< 400ml with symptoms in rest or during the walk test, the effusion will be drained and examinations will be repeated. In case of pericardial effusion of predefined size and location, either the surgeon on call or a cardiologist will be consulted.
  Interventions: Procedure: pleuracentesis

INTERVENTIONS:
Procedure: pleuracentesis — Direct needle drainage of pleural effusions with dynamic ultrasound technique
  Arms: pleuracentesis

SUMMARY:
One of the most common postoperative complications after open cardiac surgery is fluid accumulation between the pleural membranes or in the pericardial sac. This study investigates the consequence of such fluid accumulations on physical performance, recovery-time, cardiac and respiratory complications, and quality of life. Half of the participants will be followed closely and offered fluid drainage at a low threshold, and half of the participants will follow the current postoperative regimen.

DETAILED DESCRIPTION:
Introduction:

Knowledge concerning the impact of pleural and pericardial effusions on physical performance, recovery-time, cardiac and respiratory complications, and quality of life after open cardiac surgery is scarce. A more aggressive approach towards effusions has been suggested, but further studies are needed.

Objectives:

1. to determine the size of pleural and pericardial effusion that results in at least 30% reduction of physical performance in the 6-minute walk test.
2. to compare the improvement in physical performance between the intervention group and the control group, measured from baseline to day 30 after surgery.

Materials and methods:

A randomised controlled intervention trial. Patients admitted for open cardiac surgery (aortic valve surgery, coronary artery bypass graft surgery and combinations) will be randomised into either an intervention group or a control group. The intervention group will be followed with physical tests and ultrasonic examination the month following surgery. Pleural or pericardial effusion of a predefined size will be drained. The control group will follow the current postoperative regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Admitted for elective aortic valve surgery, coronary artery bypass graft surgery or combinations.
* Be able to understand the written and oral patient information and to give informed consent.

Exclusion Criteria:

* Surgical combinations involving the mitral valve since they are already examined with full echocardiography prior to discharge, which may influence protocol driven decisions.
* Simultaneous participation in any other clinical intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
change in walking distance before and after intervention | day 4, day 15, day 30
  The primary outcome measure is the change in walking distance before and after pleuracentesis, subsequently the size of pleural effusion (both cm measured on ultrasound and drained volume) that results in a reduction of distance in the 6 minute walk test of at least 30%.

SECONDARY OUTCOMES:
change in walking distance from baseline to day 30 after surgery | day 0 and day 30
  The difference in walking distance from before surgery (day 0) to after surgery (day 30) will be compared between the intervention arm (+ pleuracentesis) and the control arm (standard postoperative regimen)

OTHER OUTCOMES:
needle pleuracentesis versus pigtail catheter | day 0, day 4, day 15 and day 30
  To asses how much of the pleural effusion is drained when performing needle puncture instead of inserting a pigtail catheter. Secondary to compare the complication rate of the two procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E. Hjortdal, MD PHD DMSc, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

REFERENCES:
- [Derived] Hansen LS, Hjortdal VE, Jakobsen CJ, Heiberg J, Maagaard M, Sloth E. Early, dedicated follow-up and treatment of pleural effusions enhance the recovery rate after open cardiac surgery: results from a randomized, clinical trial. Eur J Cardiothorac Surg. 2017 Jan;51(1):58-66. doi: 10.1093/ejcts/ezw233. Epub 2016 Jul 11. PMID 27401709